CLINICAL TRIAL: NCT05036239
Title: Recovery After Exercise-Induced Muscle Damage
Brief Title: Recovery From 50 Eccentric Biceps Curls in Young, Untrained Men and Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian School of Sport Sciences (Other)
Collaborators: Université de Nantes (Other); Oslo University Hospital (Other); University of Oslo (Other); Syddansk Universitet, Denmark (Unknown); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Truls Raastad, Professor, Norwegian School of Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: EIMD19
Record Dates: First submitted 2021-05-10; First posted 2021-09-05 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Recovery; Muscle Damage; Muscle Stiffness; Cell Structure Alteration; Calcium Cycling

STUDY DESIGN:
Intervention Model Description: Participants perform one bout of eccentric exercise with one arm, while the contralateral arm serves as control. Which arm who receives eccentric exercise is randomized between dominant/non-dominant arm.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercised (Experimental): One bout of 50 eccentric biceps curls
  Interventions: Other: Eccentric biceps curls
- Control (No Intervention): No eccentric biceps curls

INTERVENTIONS:
Other: Eccentric biceps curls — 10 x 5 repetitions of eccentric biceps curls, interspaced by 30 seconds of rest.
  Arms: Exercised

SUMMARY:
The purpose of the study is to investigate muscle stiffness in relation to muscle damaging work and to investigate how well the change in muscle stiffness correlates with the degree of muscle damage (myofibrillar disruption and necrosis). To date, the reduction in force-generating capacity is the best non-invasive marker of muscle damage. It is already established that muscle stiffness correlates well with the decline in force-generating capacity after damaging exercise. However, the correlation between degree of muscle damage and muscle stiffness has not yet been investigated. The main focus of the study is therefore to investigate the relationship between muscle stiffness and muscle damage. Further, the researchers aim to investigate how calcium cycling is affected by damaging work, and if impaired calcium cycling may partially explain the observed reduction in force-generating capacity.

DETAILED DESCRIPTION:
Regardless of whether an individual is in rehabilitation or exercise for general health or athletic performance, resistance exercise is an essential form of exercise when the goal is to increase muscle mass, strength and function. Although, resistance exercise primarily is associated with positive effects it may also result in muscle damage when the exercise is of high intensity and/or unaccustomed. This is known as exercise-induced muscle damage (EIMD) and is reflected by a substantial decrease in force-generating capacity and often accompanied by intracellular swelling and delayed onset muscle soreness. On a cellular level, EIMD include myofibrillar disruption, inflammatory response and in severe cases of EIMD; myofibre necrosis. While EIMD with its symptoms clearly is evident, its underlying mechanisms are still to be fully elaborated.

One interesting hypothesis regarding the molecular basis of decreased muscle strength as a result of EIMD, is related to the strain of this exercise mode causing "popped" sarcomeres. When sarcomeres are stretched beyond actin-myosin overlap, some sarcomeres may over-stretch. This results in overload of membranes, leading to opening of stretch-activated channels, and subsequently influx of Ca2+. High levels of cytoplasmic Ca2+ may cause degradation of contractile proteins or Excitation-Contraction coupling proteins mediated through increased calpain activity. However, a recent study by Cully and colleagues (2017) suggest a protective mechanism post heavy-load strength training related to Ca2+-handling. Cully et al. observed formation of vacuoles in longitudinally connecting tubules post exercise when exposing fibers to 1.3 μM [Ca2+] in the cytoplasma. These vacuoles provide an enclosed compartment where Ca2+ can be accumulated, preventing Ca2+ from initiating damage to the muscle. The role of Ca2+-regulation in recovery of muscle function warrants further investigation and clarification.

To the best of the investigators knowledge, the most valid method for estimating EIMD is by investigating myofibrillar disruption, and in some cases necrosis, in muscle biopsies. This requires many resources and is rather expensive. Currently, the best non-invasive marker of muscle damage is the force deficit observed at 48 hours post exercise. However, a measurement estimating muscle damage immediately post exercise is warranted because force deficit immediately post exercise will be confounded by muscle fatigue.

A novel study performed by Lacourpaille et al. (2017) showed a strong negative correlation (-0.80) between stiffness of the muscle tissue, shear modulus, measured 30 minutes post exercise and peak isometric force measured at 48 hours post exercise and therefore a strong relationship between the decline in force production capacity and increased stiffness post exercise, suggesting a possible method to predict EIMD immediately after exercise. However, direct evidence of this association is warranted, with measurements of shear modulus and EIMD biomarkers, such as the proportion of disrupted fibers and sarcoplasmic Ca2+ regulation.

The ability to predict EIMD after training is of great interest to athletes, but also patients suffering from e.g. muscular dystrophies. Being able to predict EIMD quickly and non-invasively after exercise will help employ optimal recovery.

The aim of this project is to investigate the link between exercise-induced muscle damage (EIMD) as changes in shear modulus by ultrasound shear wave elastography, and muscle damage as observed in the analysis of muscle biopsies. The hypothesis is that there is a strong relationship between muscle stiffness acute post exercise and degree of muscle damage observed in muscle biopsies. A secondary aim is to further the understanding of cellular mechanisms causing EIMD and the role of Ca2+ in the recovery of muscle function.

ELIGIBILITY:
Inclusion Criteria:

- 18 to 35 years of age

Exclusion Criteria:

* Injury to the muscle-skeletal system
* Other conditions causing inability to perform heavy-load resistance exercise
* Having engaged in resistance exercise targeting the m. biceps brachii once a week or more over the past year

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2019-12-03 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Change in muscle strength | Baseline, and 5 minutes, 3 hours, 24 hours, 48 hours, 72 hours, and 96 hours after eccentric biceps curls
  Recovery of arm flexion torque
Change in muscle stiffness | Baseline, and 50 minutes, 3 hours, 24 hours, 48 hours, 72 hours, and 96 hours after eccentric biceps curls
  Muscle stiffness measured with shear wave elastography as mean young modulus in different conditions (static and dynamic)
Change in muscle damage | 2 hours, 48 hours, and 96 hours after eccentric biceps curls
  Development of myofibrillar disruption and necrosis observed in skeletal muscle biopsies with electron and confocal microscopy
Change in calcium cycling | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Calcium cycling in muscle single fibers and Sarcoplasmic reticulum-homogenate

SECONDARY OUTCOMES:
Change in organization of the tubular system in skeletal muscle | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Quantification of transverse and longitudinal tubules, and number of Vacuoles in single fibers using confocal microscopy

OTHER OUTCOMES:
Change in HSP70 | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Localization of HSP70 in skeletal muscle using Western blotting
Change in AlphaB-crystallin | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Localization of alphaB-crystallin in skeletal muscle using Western blotting
Change in Fiber-specific AlphaB-crystallin staining intensity | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Change in staining intensity of AlphaB-crystallin in type-I and type-II skeletal muscle fibers using Immunohistochemistry
Change in Fiber-specific HSP70 staining intensity | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Change in staining intensity of HSP70 in type-I and type-II skeletal muscle using Immunohistochemistry
Change in Fatigue | Baseline and 1 hour after eccentric biceps curls
  Electrical stimulation of m. biceps brachii at 20 and 50 Hz
Change in Muscle soreness | Baseline, 15 minutes, 23 hours, 47 hours, 71 hours, and 95 hours after eccentric biceps curls
  Subjective rating of muscle soreness using a VAS-scale (0-10)
Change in Muscle swelling (circumference) | Baseline, 15 minutes, 23 hours, 47 hours, 71 hours, and 95 hours after eccentric biceps curls
  Circumference of upper arm measured 2 cm above humeral epicondyles and midbelly of m. biceps brachii
Change in Muscle swelling (thickness) | Baseline, 2 minutes, 23 hours, 47 hours, 71 hours, and 95 hours after eccentric biceps curls
  Thickness at midbelly of m. biceps brachii using ultrasound B-mode
Change in Creatine kinase | Baseline, 2,5 hours, 24 hours, 48 hours, 72 hours, and 96 hours after eccentric biceps curls
  Level of serum creatine kinase
Change in Myoglobin | Baseline, 2,5 hours, 24 hours, 48 hours, 72 hours, and 96 hours after eccentric biceps curls
  Level of serum myoglobin
Change in Titin | Baseline, 2,5 hours, morning day 2, morning day 3, morning day 4, and morning day 5 after eccentric biceps curls
  Level of titin-N fragment in urine
Change in Troponin I | Baseline, 2,5 hours, 24 hours, 48 hours, 72 hours, and 96 hours after eccentric biceps curls
  Level of serum Troponin I in fast and slow twitch muscle fibers
Change in Macrophage infiltration | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Presence of macrophages in skeletal muscle using Immunohistochemistry
Muscle fiber type | 2 hours after eccentric biceps curls
  Fiber type composition in cross-sections of muscle samples using Immunohistochemistry
Muscle fiber type | 48 hours after eccentric biceps curls
  Fiber type composition in cross-sections of muscle samples using Immunohistochemistry
Muscle fiber type | 96 hours after eccentric biceps curls
  Fiber type composition in cross-sections of muscle samples using Immunohistochemistry
Change in Calcium-related protein abundances in skeletal muscle | 2 hours, 48 hours and 96 hours after eccentric biceps curls
  Levels of proteins and phosphorylation status using Western blotting

CONTACTS AND LOCATIONS:
Overall Officials: Truls Raastad, PhD, Principal Investigator — Norwegian School of Sport Sciences
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No